CLINICAL TRIAL: NCT07387354
Title: A Phase 1/2 Study of Pacritinib in Combination With Azacitidine for the Treatment of IPSS-M Moderate Low to Very High Risk Myelodysplastic Syndrome
Brief Title: Pacritinib With Aza for Upfront Myelodysplastic Syndrome
Acronym: MDS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iRIS ID- 2024-2998; JT 36125 (Other: JeffTrial Number)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes; MDS; Myelodysplastic Syndrome, Unclassifiable; Hematologic Diseases; Bone Marrow Disease; Myeloproliferative Neoplasm
Keywords: Pacritinib; Azacitidine; IPSS-M; JAK/STAT; JAK/IRAK1; NF-κβ; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Hematologic Diseases; Bone Marrow Diseases; Myeloproliferative Disorders | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Azacitidine; Bone Marrow Examination; Clinical Laboratory Techniques; Electrocardiography; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pacritinib 100 mg twice daily (200 mg total) - Dose level X-1 + azacitidine (Experimental): Participants will receive oral Pacritinib 100mg administered twice daily (200 mg total) in combination with Azacitidine 75mg/m² administered intravenously or subcutaneously on Days 1-7 of each 28-day cycle. The Phase 1 portion uses a 3+3 dose-escalation design to identify the recommended Phase 2 dose (RP2D)
  Interventions: Drug: Pacritinib; Drug: Azacitidine; Procedure: Bone Marrow Biopsy and Aspirate; Diagnostic Test: Laboratory Testing; Diagnostic Test: Electrocardiogram; Other: Quality of Life in Myelodysplasia Scale
- Pacritinib 100 mg AM / 200 mg PM (300 mg total) - Dose level X (starting dose) + azacitidine (Experimental): Participants will receive oral Pacritinib administered twice daily in combination with Azacitidine administered intravenously or subcutaneously on Days 1-7 of each 28-day cycle. The Phase 1 portion uses a 3+3 dose-escalation design to identify the recommended Phase 2 dose (RP2D); the Phase 2 portion uses a Simon two-stage design to evaluate efficacy and safety at the RP2D.
  Interventions: Drug: Pacritinib; Drug: Azacitidine; Procedure: Bone Marrow Biopsy and Aspirate; Diagnostic Test: Laboratory Testing; Diagnostic Test: Electrocardiogram; Other: Quality of Life in Myelodysplasia Scale
- Pacritinib 200 mg twice daily (400 mg total) - Dose level X+1 + azacitidine (Experimental): Participants will receive oral Pacritinib administered twice daily in combination with Azacitidine administered intravenously or subcutaneously on Days 1-7 of each 28-day cycle. The Phase 1 portion uses a 3+3 dose-escalation design to identify the recommended Phase 2 dose (RP2D); the Phase 2 portion uses a Simon two-stage design to evaluate efficacy and safety at the RP2D.
  Interventions: Drug: Pacritinib; Drug: Azacitidine; Procedure: Bone Marrow Biopsy and Aspirate; Diagnostic Test: Laboratory Testing; Diagnostic Test: Electrocardiogram; Other: Quality of Life in Myelodysplasia Scale
- Pacritinib RP2D + azacitidine - Phase 2 Expansion (Experimental): Participants receive Pacritinib at the recommended Phase 2 dose (RP2D) as determined during the Phase 1 dose-escalation portion of the study, in combination with Azacitidine 75 mg/m2 intravenously or subcutaneously on Days 1-7 of each 28-day cycle.
  Interventions: Drug: Pacritinib; Drug: Azacitidine; Procedure: Bone Marrow Biopsy and Aspirate; Diagnostic Test: Laboratory Testing; Diagnostic Test: Electrocardiogram; Other: Quality of Life in Myelodysplasia Scale

INTERVENTIONS:
Drug: Pacritinib — Pacritinib is an oral kinase inhibitor with activity against wild-type JAK2, mutant JAK2V617F, FLT3, IRAK1, and ACVR1. Administered twice daily at 200mg or 400mg total daily dose per Phase 1 dose escalatio
  Other Names: Vonjo
Drug: Azacitidine — Lyophilized powder in 100mg single dose vials to be diluted in saline to generate 75 mg/m2 intravenous or subcutaneous solutions. Azacitidine to be given at 75mg/m2 infusion days 1-7 every four weeks.
  Other Names: Vidaza; 5-Azacytidine
Procedure: Bone Marrow Biopsy and Aspirate — Bone marrow aspiration and biopsy as per standard of care obtained at baseline, infusion visit Days 2-7, and study completion Day 112.
  Other Names: BMA/BMB; Bone Marrow Examination; Bone Marrow Test
Diagnostic Test: Laboratory Testing — Laboratory Tests to include CMP, Magnesium Phosphorous, LDH, Uric Acid, and CBC with Differential will be performed at baseline, Cycle 1, and at the start of each subsequent cycle.
  Other Names: CMP; Magnesium Phosphorous; LDH; Uric Acid
Diagnostic Test: Electrocardiogram — ECG will be obtained on day 7 of each cycle to document QTc interval. ECGs will be performed at clinician's discretion in addition to ones required by study as outlined above.
  Other Names: ECG
Other: Quality of Life in Myelodysplasia Scale — Quality of life will be assessed using QUALMS at baseline and after completion of 4 cycles (Day 112). QUALMS is a 38-item assessment tool for patients with myelodysplastic syndromes (MDS).
  Other Names: QUALMS

SUMMARY:
This study will be conducted as a phase 1/2 study of safety and preliminary efficacy of pacritinib in combination with azacitidine for IPSS-M moderate low to very high risk MDS. Phase one will be a 3 + 3 design to assess the dose for the phase two portion. The phase two portion will employ a simon min-max two-stage design whereby fifteen patients will be enrolled in the first stage then ten more if at least two patients in stage one have a response. The dosing of pacritinib for the phase two study will be based on the phase one findings. Standard dosing of azacitidine will be used. A correlative study will be conducted in conjunction with the trial where we will measure whole blood collected pre-treatment and at four days post-treatment to measure intracellular flow and phosflow to detect JAK/STAT, NF-κβ, and AKT/mTOR signaling in patient samples and how treatment affects these pathways.

DETAILED DESCRIPTION:
Phase I Design:

Phase one will be a 3 + 3 design to assess the dose for the phase two portion. We will use a two-stage accrual design at each dose considered. We will initially enter three subjects at 300mg total. If none of the three experiences a dose-limiting toxicity (DLT) we will proceed to 400mg total as our second dose. If one of the three experiences DLT, we will enter three additional patients at 300mg total. If at most one experience DLT in the cohort of six at 300mg total, we will proceed with 400mg total as our second dose. If two or more experience DLT in the cohort of six at 300mg total, we will proceed to 200mg total as our second dose. If two or more experiences DLT in the original cohort of three at 300mg total, we will proceed to 200mg total as our second dose.

For the second dose (400mg or 200mg) three subjects will be initially treated. If none or one of the three experience a DLT, then we will accrue three more subjects at that dose. If at most one of six experience a DLT, then the second dose will be given for phase two, called the highest tested dose if 400mg and highest tolerated dose if 200mg. If two or more of six experience a DLT on 400mg total, then the previous dose (300mg total) will be declared the highest tolerated dose. If two or more of six experience a DLT on 200mg total, then we will terminate the trial.

If there are two or more dose-limiting toxicities in the cohort of three on 400mg total, then the previous dose (300mg total) will be declared highest tolerated dose. If there are two or more dose-limiting toxicities in the cohort of three on 200mg total, then we will terminate the trial.

No patient will be treated at a higher dose until the three or six patients have completed their toxicity evaluation period at the current dose. With this plan, a dose with a 50% or greater probability of causing a dose-limiting toxicity has at most a 12.5% chance of satisfying the conditions for dose escalation after the first three subjects and at least a 50% chance of stopping at three. With the two-stages (3-6) together, there is at most a 17.2% chance of escalation.

Phase II Design:

Phase two of this trial is designed with the potential for early termination in the case of failure to prove efficacy. The design will be a Simon's two-stage admissible minimax design.40 Choice of design is guided by a desire to stop the trial early if the actual ORR rate is 10% or less. If the ORR rate is 30% or greater, we would like to have a low probability of failing to conclude effective.

With this design, we have no more than a 10% chance of concluding ineffective (≤10% ORR) when the ORR is at least 30%. Similarly, we have no more than a 5% chance of concluding effective (≥30% ORR) when it is ineffective. If the actual ORR is 10% or lower, we have 55% probability that the trial will stop after the first fifteen subjects. The first stage of fifteen patients will include the patients in the phase one portion who were on the chosen phase two dose. If there are greater than five successes after the total twenty-five patient cohort, then the trial is considered a success.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following inclusion criteria to be eligible to participate in the study:

  1. Patients must have histologic evidence of intermediate to high-risk myelodysplastic syndrome defined as having an IPSS-M score of moderate low, moderate high, high or very high risk. This will be assessed based on evaluations performed prior to screening for trial. Of note, the most recent evaluation pre-trial may be used which does not have to necessarily be at diagnosis.
  2. Subjects must have recovered from the toxic effects of any prior chemotherapy to ≤ Grade 1 (except alopecia).
  3. Required screening visit laboratory values: CrCL ≥45; total bilirubin <2xULN except for patients with known Gilbert's disease; SGPT (ALT) ≤2xULN, PTT ≤1.5xULN.
  4. Negative pregnancy test for women with child-bearing potential at screening visit.
  5. Initial screening baseline QTc ≤480ms.
  6. Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
  7. Patients must have an absolute neutrophil count of ≥750 to enroll in study, this must be achieved without the addition of growth factor medication.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Any prior exposure to a hypomethylating agent (azacitidine or decitabine)
  2. Any prior exposure to JAK2 inhibitor therapy (ie ruxolitinib or prior pacritinib therapy)
  3. Any exposure within the past seven days of initiation of study treatment to a strong CYP3A inhibitor/inducer.
  4. Subjects must not be receiving any chemotherapy agents (except hydroxyurea) within the past thirty days.
  5. Subjects must not be receiving growth factors (erythropoietin mimetics, granulocyte stimulating factor mimetics, thrombopoietin mimetics) for two weeks prior to enrollment bone marrow. Subjects may not receive growth factors for the duration of this study.
  6. Subjects with a "currently active" second malignancy, other than curatively treated non-melanoma skin cancer, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pT2 with Gleason Score ≤ 6 and postoperative PSA <0.5 ng/mL), or other adequately treated carcinoma-in-situ are eligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 1 year.
  7. Subjects with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure (NYHA class 2), myocardial infarction within the past 6 months or serious uncontrolled cardiac arrhythmia are not eligible.
  8. Bleeding event grade >=2 (CTCAE 5.0) within prior three months unless provoked (e.g., by surgery or trauma)
  9. Use of anticoagulant or antiplatelet agents within fourteen days prior to day one with the exception of low dose aspirin (81mg daily).
  10. Subjects with other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study are ineligible.
  11. Active or uncontrolled diarrhea or constipation.
  12. Subjects must not have evidence of active disease in the CNS.
  13. Subjects must not have received any investigational agents within fourteen days or five half-lives (whichever is longer) of study entry.
  14. Subjects must not be pregnant or breastfeeding. Pregnancy tests must be obtained for all females of child-bearing potential. Pregnant or lactating patients are ineligible for this study due to the unknown human fetal or teratogenic toxicities of pacritinib. Males or women of childbearing potential may not participate unless they have agreed to use a highly effective contraceptive method (defined in section 10.4.4).
  15. Subjects who have uncontrolled infection are not eligible. Patients must have any active infections under control. Fungal disease must be stable for at least two weeks before study entry.
  16. Subjects with bacteremia must have documented negative blood cultures prior to study entry.
  17. Subjects who are currently candidates for allogeneic transplantation, have a suitable donor, and are willing to undergo transplantation prior to study start.
  18. Subjects who cannot hold a medication, over the counter, or supplemental product that in the investigator's opinion may put the patient at increased harm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Optimal Dose of Pacritinib in Combination with Azacitidine - Phase 1 | Baseline through Day 28 (Cycle 1)
  "Phase 1 of the study is designed to determine the optimal dose of pacritinib in combination with azacitidine in subjects with moderate, high, and very high risk MDS.
  The optimal dose (recommended Phase 2 dose, RP2D) will be defined as the highest dose level associated with an acceptable rate of dose-limiting toxicities (DLTs) during Cycle 1, using a standard 3 + 3 dose-escalation design.
  DLTs are defined per NCI CTCAE v5.0 (Section 7.5 of protocol):
  * Any grade ≥ 3 non-hematologic toxicity (excluding grade 3 nausea, vomiting, or diarrhea that improves to ≤ grade 2 within 5 days);
  * Prolonged grade 4 hematologic toxicities not due to persistent disease;
  * Any grade 5 toxicity not attributable to disease progression. Safety, tolerability, and pharmacodynamic data will support RP2D selection. "
Rate of Dose Limiting Toxicities (DLTs) - Phase 1 | Baseline through Day 28 (Cycle 1)
  "the proportion of participants experiencing dose limiting toxicities (DLTs) occurring within thirty days of first dose of study agent that meets the following qualifications and is potentially related to study medication or combination will be considered a dose limiting toxicity. DLTs are defined per NCI CTCAE v5.0 as:
  * Any grade ≥ 3 non-hematologic toxicity (excluding grade 3 nausea, vomiting, or diarrhea that improves to ≤ grade 2 within 5 days);
  * Prolonged grade 4 hematologic toxicities (e.g., neutropenia or thrombocytopenia not due to persistent disease);
  * Any grade 5 toxicity not attributable to disease progression."
Overall Response Rate (ORR) - Phase 2 | Baseline through Week 16 (approximately 4 months)
  Overall response rate (ORR) = patients achieving CR (or CR equivalent), PR, CRL, CRh, or hematologic improvement (HI) ÷ total patients. ORR per IWG 2023 criteria; hematologic response per IWG 2018. Responses: CR, CR equivalent, PR, CRL, CRh, or HI (erythroid, platelet, neutrophil).
  IWG 2023:
  CR: BM <5% blasts; Hb ≥10 g/dL; platelets ≥100×10⁹/L; ANC ≥1.0×10⁹/L; no blood blasts.
  CR equivalent: Baseline <5% blasts + complete cytogenetic response. PR: CR criteria except ≥50% blast reduction (still ≥5%). CRL: <5% blasts; no blood blasts; recovery of 1-2 lineages. CRh: <5% blasts; no blood blasts; platelets >50×10⁹/L; ANC >0.5×10⁹/L.
  IWG 2018 HI:
  HI-E: Hb ↑ ≥1.5 g/dL or RBC TI ≥8 wks. HI-P: Platelets ↑ ≥30×10⁹/L or from <20 to >20×10⁹/L + ≥100% ↑. HI-N: ≥100% ↑ and absolute ↑ ≥0.5×10⁹/L.

SECONDARY OUTCOMES:
Duration of Overall Response Rate - Phase 2 | Up to 2 years after last patient enrolled
  Time from first documented response (CR, PR, or HI per IWG criteria) until relapse, progression, or death from any cause.
Overall Surival - Phase 2 | Up to 24 months
  Time from study enrollment to death from any cause.
Number of Treatment Emergent Adverse Events (TEAEs) | Baseline through Cycle 4, plus 30 days (Approximately 5 months)
  Incidence, seriousness, severity, outcome, discontinuation or dose modifications related to TEAEs. This is separate from the primary endpoint of phase one which will be rate of DLTs.
Molecular Response Rate (Phase 2) | Baseline through Week 16 (approximately 4 months)
  Assessment of molecular response will be done via rate of disappearance of relevant mutations via next-generation sequencing on pre and post treatment bone marrow samples.
Change in Intracellular Signaling Pathway Activation (JAK/STAT, NF-κB and AKT/mTOR | Baseline
  Whole blood along with bone marrow aspirate with be collected pre and post treatment to assess intracellular flow and phosflow to detect NF-κB, JAK/STAT, and AKT/mTOR signaling within all myeloid cells. Post treatment will be compared to pre-treatment for all flow markers (intra- and extracellular) for changes in signaling and WBC maturation. Patient genetics will also be evaluated in the context of signaling response and maturation
Change in Intracellular Signaling Pathway Activation (JAK/STAT, NF-κB and AKT/mTOR | After four days of azacitidine and pacritinib therapy
  Whole blood along with bone marrow aspirate with be collected pre and post treatment to assess intracellular flow and phosflow to detect NF-κB, JAK/STAT, and AKT/mTOR signaling within all myeloid cells. Post treatment will be compared to pre-treatment for all flow markers (intra- and extracellular) for changes in signaling and WBC maturation. Patient genetics will also be evaluated in the context of signaling response and maturation
Assessment of Quality of Life Using the quality of life in myelodysplasia scale (QUALMS) | At Baseline
  To measure quality of life pre-treatment and after four cycles of treatment using the quality of life in myelodysplasia scale (QUALMS). The Quality of Life in Myelodysplasia Scale (QUALMS) is a 38-item, disease-specific questionnaire used to measure the health-related quality of life in patients with myelodysplastic syndromes (MDS). It includes three subscales for physical burden, emotional burden, and benefit finding, and a total score ranges from 0 to 100, where a higher score indicates a better quality of life.
Assessment of Quality of Life Using the quality of life in myelodysplasia scale (QUALMS) | After 4 cycles of treatment (approximately 112 days)
  To measure quality of life pre-treatment and after four cycles of treatment using the quality of life in myelodysplasia scale (QUALMS). The Quality of Life in Myelodysplasia Scale (QUALMS) is a 38-item, disease-specific questionnaire used to measure the health-related quality of life in patients with myelodysplastic syndromes (MDS). It includes three subscales for physical burden, emotional burden, and benefit finding, and a total score ranges from 0 to 100, where a higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chetan Jeurkar, DO, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University